CLINICAL TRIAL: NCT02328365
Title: Screening and Systematic Follow-up for Cardiopulmonary Comorbidity in Patients Having Surgery for Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Comorbidity
Record Dates: First submitted 2014-12-10; First posted 2014-12-31 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Comorbidity; Perioperative Care; Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (No Intervention): Patients screened positive for cardiopulmonary disease and having a medical (pulmonary and/or cardiology) visit preoperatively, but randomized to standard follow-up
- Intervention (Experimental): Patients screened positive for cardiopulmonary disease and having a medical (pulmonary and/or cardiology) visit preoperatively, but randomized to structured medical follow-up after operation
  Interventions: Other: Structured medical follow-up after operation

INTERVENTIONS:
Other: Structured medical follow-up after operation — Patients in the intervention arm are seen by a physician on the 4th or 5th postoperative day before discharge to pick up and manage any medical problems, and are furthermore seen in the cardiology clinic 1 month after operation, and in the pulmonary medicine clinic 1 and 3 months after operation
  Arms: Intervention

SUMMARY:
More than one third of patients with colorectal cancer (CRC) suffer from comorbidity such as heart and lung diseases. This comorbidity markedly impairs survival after surgical treatment owing to increased mortality within the first weeks to months after surgery. Since the operation itself constitutes a severe challenge to the patient's cardiopulmonary system, this study aims to elucidate whether a more systematic perioperative management and follow-up of colorectal cancer patients with cardiopulmonary comorbidity may improve their outcome as measured by complications, hospitalisation times, and survival.

DETAILED DESCRIPTION:
Background and overview

More than one third of patients with colorectal cancer (CRC) suffer from comorbidity such as heart and lung diseases. This comorbidity markedly impairs survival after surgical treatment owing to increased mortality within the first weeks to months after surgery, and this increased mortality is related to medical complications such as heart and lung complications. Since the operation itself constitutes a severe challenge to the patient's cardiopulmonary system, this study aims to elucidate whether a more systematic perioperative management and follow-up of colorectal cancer patients with cardiopulmonary comorbidity may improve their outcome as measured by complications, hospitalisation times, and survival within the first year.

All patients scheduled for elective surgical treatment of colorectal cancer at Vejle Hospital are screened by a study nurse for cardiopulmonary comorbidity to determine their eligibility for inclusion. If they fulfil inclusion criteria, they are seen preoperatively by a cardiologist and/or a pulmonary physician and undergo echocardiography and/or spirometry.

Included patients are randomized postoperatively to either standard follow-up alone ("standard" group) or standard follow-up supplemented with structured medical management and follow-up ("intervention" group). Patients in the intervention group are examined on the 4th or 5th postoperative day by an experienced physician from the Department of Internal Medicine. Furthermore, the intervention group is followed up at outpatient visits 1 and 3 months postoperatively. The 1-month visit includes a cardiology visit with echocardiography and ECG, and a pulmonary medicine visit with spirometry. The 3-month visit includes only a pulmonary medicine visit with spirometry.

Mortality, cardiopulmonary complications, hospitalisation time and treatment changes induced by the structured follow-up will be recorded as outcome measures for the intervention.

Hypothesis

Patients with cardiopulmonary comorbidity who have their standard follow-up extended to include a structured medical management and follow-up after surgery for colorectal cancer obtain a better outcome as measured by less cardiopulmonary morbidity and better survival within the first year.

Aim

To test a study design with systematic preoperative screening for cardiopulmonary comorbidity and postoperative randomization of eligible patients to either standard followup alone or standard follow-up supplemented with structured medical management and follow-up after operation for colorectal cancer.

Design

A randomized feasibility study. Based on older data, it will require approximately 400 patients in each arm to demonstrate a 10 % reduction in the expected mortality. This study aims to test the design and acquire more reliable mortality data in each arm in order to establish the basis for a larger multicentre study.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for elective surgical treatment of colorectal cancer at Vejle Hospital

Exclusion Criteria:

* Patients younger than 18 years, patients who are not legally competent, and patients with disseminated cancer and limited life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Postoperative mortality at one year | One year

SECONDARY OUTCOMES:
Short-term postoperative mortality | 30 days and 6 months
Medical complications | 3 months
  Incidence of postoperative medical complications as classified in the Danish national bowel cancer database (stroke, ACS, aspiration, pneumonia, heart failure, arrhythmia, pulmonary embolism, lung failure, renal failure, sepsis, deep vein thrombosis, arterial embolism, other) and graded according to Clavien. Particular focus on cardiopulmonary complications

OTHER OUTCOMES:
Hospitalization time | 30 days
Readmissions | 3 months
Findings and interventions at medical visits | 3 months
  Incidence of intercurrent or present medical complications as described in Outcome 3. Judgement whether the complication was 1. already identified and optimally managed by others, 2. identified but not optimally managed, or 3. was undisclosed until the medical visit. Any interventions by the visiting physician graded (no intervention, change in medication, unplanned outpatient visit, admission to hospital as inpatient)

CONTACTS AND LOCATIONS:
Overall Officials: Hans B Rahr, MD DMSc, Study Chair — Department of Surgery
Locations (1):
- Vejle Hospital, Department of Surgery, Vejle, Denmark

REFERENCES:
- [Derived] Rahr HB, Streym S, Kryh-Jensen CG, Hougaard HT, Knudsen AS, Kristensen SH, Ejlersen E. Screening and systematic follow-up for cardiopulmonary comorbidity in elective surgery for colorectal cancer: a randomised feasibility study. World J Surg Oncol. 2019 Jul 22;17(1):127. doi: 10.1186/s12957-019-1668-7. PMID 31331339